CLINICAL TRIAL: NCT00969527
Title: Assessment of the Efficacy of Oncoxin+Viusid Administration in the Treatment of Rheumatoid Arthritis
Brief Title: Efficacy of Oncoxin Plus Viusid in the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Juan Carlos Delgado Morales, "Fructuoso Rodríguez" Orthopedic Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-0903-CU
Record Dates: First submitted 2009-08-27; First posted 2009-09-01 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Oncoxin; Viusid; dietary supplements; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Viusid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Oncoxin + Viusid
  Interventions: Dietary Supplement: Oncoxin + Viusid
- B (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oncoxin + Viusid — 50 ml of Oncoxin + Viusid (Orally administered) twice a day, for 12 weeks.
  Arms: A
Dietary Supplement: Placebo — 50 ml of Placebo (orally administered) twice a day, for 12 weeks.
  Arms: B

SUMMARY:
The purpose of the study is to assess the efficacy of Oncoxin+Viusid administration in the treatment of rheumatoid arthritis. The duration of this double-blind placebo controlled phase 3 clinical trial will be 12 weeks. The estimated number of persons with rheumatoid arthritis to be recruited and randomized for the study is 86. The primary outcome measure: DAS28 score will be assessed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive subjects with recent onset rheumatoid arthritis
* Signed informed consent

Exclusion Criteria:

* Subjects with rheumatoid arthritis symptoms other than those associated with joints at disease onset
* Subjects with joint function impairment secondary to other conditions not associated with rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score (DAS 28 score) at week 12. | 12 weeks
  DAS 28=(0.56√NAD+ 0.28√NAT+0.7ln⁡VSG+0.14EGE) where NAD: number of joints with pain; NAT: number of joints with increased volume; VSG: sedimentation rate of erythrocytes; EGE: Global assessment of disease by the patient on a visual analog scale (1 to 100 mm)

SECONDARY OUTCOMES:
Number of patients with Adverse Events at week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Delgado Morales, MD, Principal Investigator — "Fructuoso Rodríguez" Orthopedic Hospital
Locations (1):
- Fructuoso Rodriguez Orthopedic Hospital, Havana, Cuba